CLINICAL TRIAL: NCT06566729
Title: Application of Molecular Residual Disease in the Recurrence Monitoring and Response Predicting of High-risk Early Breast Cancer
Brief Title: MRD in High-risk EBC
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Ruijin Hospital
Other Study IDs: RJBC2301
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: MRD; breast cancer; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Peripheral blood sample collection — In this study, peripheral blood samples would be collected before adjuvant chemotherapy, after adjuvant chemotherapy and every 3 months thereafter until 2 years after surgery.

SUMMARY:
This study is a multicenter, prospective, observational cohort study, 125 patients with early-stage high-risk breast cancer will be enrolled, perioperative surgical specimens, peripheral blood specimens before and after adjuvant therapy and follow-up will be collected, and the predictive effect of MRD of molecular residual lesions on recurrence events and drug efficacy will be evaluated through dynamic monitoring, so as to further accurately stratify the risk and guide clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Age ≥18 years old
* Undergoing breast surgery, the surgical specimen was diagnosed as invasive breast cancer by the central laboratory and met any of the following conditions:

  1. Hormone receptor-positive/HER2-negative breast cancer, the number of lymph node metastases ≥ 4;
  2. HER2-positive breast cancer, lymph node metastasis≥4;
  3. Triple negative breast cancer, the number of lymph node metastases ≥ 1;
* ECOG 0-1
* Willing to cooperate in clinical research-related treatment and follow-up, with good patient compliance

Exclusion Criteria:

* Confirmed distant metastases site
* History of other malignancy
* Psychopaths or other reasons unable to comply with treatment
* Concomitant uncontrolled lung disease, severe liver and kidney disease, severe infection, active peptic ulcer requiring treatment, coagulation disorders, connective tissue disease, or bone marrow suppression, and cannot tolerate chemotherapy and other related treatments
* HIV carrier or HBC/HCV infected
* Current or recent (within 30 days prior to enrollment) use of participation in another investigational program or use of another investigational drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Hormone receptor-positive/HER2-negative breast cancer, the number of lymph node metastases ≥ 4;
  2. HER2-positive breast cancer, lymph node metastasis≥4;
  3. Triple negative breast cancer, the number of lymph node metastases ≥ 1;
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | 5 years after surgery
  Defined as the time from the diagnosis of the disease to the first occurrence of a local recurrence of breast cancer, distant recurrence, or death from any cause

SECONDARY OUTCOMES:
Overall survival | 5 years after surgery
  Defined as the time from the diagnosis of the disease to the first occurrence of a death event from any cause
Lead time | 2 years after surgery
  Defined as the time from the first positive peripheral blood MRD test to radiologically confirmed metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No